CLINICAL TRIAL: NCT01828476
Title: A Phase II Study of ABT-263/Abiraterone (Arm A) or ABT-263/Abiraterone and Hydroxychloroquine (Arm B) in Patients With Metastatic Castrate Refractory Prostate Cancer (CRPC) and Progression Following Chemotherapy and Abiraterone
Brief Title: Navitoclax and Abiraterone Acetate With or Without Hydroxychloroquine in Treating Patients With Progressive Metastatic Castrate Refractory Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Investigator left the organization.
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other); National Cancer Institute (NCI) (NIH); AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 081214; Pro2013002775 (Other: Rutgers IRB #); P30CA072720 (NIH); NCI-2013-02403 (Other: NCI Trial ID)
Record Dates: First submitted 2013-03-26; First posted 2013-04-10 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; hormone-resistant prostate cancer; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; navitoclax; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM A (Experimental): Abiraterone with ABT-263
  Interventions: Drug: Abiraterone; Drug: ABT-263
- ARM B (Experimental): Abiraterone with both ABT-263 and Hydroxychloroquine
  Interventions: Drug: Abiraterone; Drug: ABT-263; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Abiraterone — ARM A(Abiraterone with ABT-263) and ARM B(Abiraterone with both ABT-263 and Hydroxychloroquine)
Drug: ABT-263 — ARM A(Abiraterone with ABT-263) and ARM B(Abiraterone with both ABT-263 and Hydroxychloroquine)
Drug: Hydroxychloroquine — ARM B(Abiraterone with both ABT-263 and Hydroxychloroquine)
  Arms: ARM B

SUMMARY:
The purpose of this study is to assess the effect of combining abiraterone with medicines that may block some of the ways that cells become resistant to abiraterone. The investigators hope that these combinations of medicines will result in prostrate cancer cells dying.

This study will see if overcoming diseases resistance to abiraterone will restore sensitivity to androgen deprivation therapy.

DETAILED DESCRIPTION:
Subjects will be either treated on one of the earlier dosing regimens or randomly assigned to one of two groups or ARMs of this study.

ARM A will receive Abiraterone with ABT-263.

ARM B will receive Abiraterone with both ABT-263 and Hydroxychloroquine

In the beginning of the study a total of 18 patients may get one of three dose levels. A total of nine (9) patients per each arm will be started at a low dose and given increasing doses if no side effects are seen. In this part of the study three patients will be enrolled at each dose level for each individual arm starting with Arm A followed by Arm B.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had evidence of disease progression while receiving primary androgen suppression therapy by orchiectomy or other primary hormonal therapy and abiraterone (Specifically, patients can have received multiple prior additional androgen axis targeting agents including enzalutamide, and prior chemotherapy, but must have had progression (as defined in 5.1.2) while receiving abiraterone either currently or in the past). Patients currently on abiraterone may continue with the start of the study drug(s).
* Patients must have evidence of disease progression during current or prior therapy with abiraterone with either:

  1. Biochemical progression as defined as rising PSA from a nadir or baseline (whichever was lowest) confirmed on a second determination at least 1 week later that must be higher than the first and must have reached ≥2ng/ml (if no other evidence of progression); or
  2. New Metastases on bone scan (at least 2); or
  3. Progression of measurable disease on CT scan by RECIST criteria
* Age >18 years and an estimated life expectancy of at least 6 months.
* Treatment with at least 2 months of abiraterone prior to progression
* ECOG performance status ≤ 2. (See Appendix A)
* Patients must be ≥ 4 weeks since completing their prior therapy (including surgery, radiation therapy or investigational therapy (including targeted small molecule agents)). All previous clinically significant treatment-related toxicities have resolved to ≤ Grade 1. Patients must be ≥ 4 weeks since prior therapy with an anti-androgen
* Adequate renal function (serum creatinine ≤ 2.0 mg/dL or creatinine clearance ≥50 ml/min)
* Total bilirubin must be within 1.5 X the normal institutional limits. If total bilirubin is outside the normal institutional limits, assess direct bilirubin. The direct bilirubin must be within normal parameters. Transaminases (SGOT and/or SGPT) must be less than 1.5X ULN concomitant with alkaline phosphatase less than 5X the ULN.
* An ANC >1500/μl, hemoglobin > 8.5 g/dl, and platelet count >100,000/mm3 are required.
* Serum testosterone (total) less than 25 ng/ml at time of enrollment.
* Bisphosphonates/RANK-ligand inhibitor allowed if started prior to study treatment
* Patient must consent to using effective contraception while on treatment and for 3 months thereafter
* Subject must voluntarily sign and date an informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures

Exclusion Criteria:

* Known infection with HIV or subject has tested positive for HIV (due to potential drug-drug interactions between anti-retroviral inhibitors and ABT-263, as well as anticipated ABT-263 mechanism based lymphopenia that may potentially increase the risk of opportunistic infections and potential drug-drug interactions with certain anti infective agents). Patients without prior HIV testing will not be required to be tested.
* Second primary malignancy except most situ carcinoma (e.g. adequately treated non-melanomatous carcinoma of the skin) or other malignancy treated at least 5 years previously with no evidence of recurrence.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

  * active systemic fungal infection;
  * diagnosis of fever and neutropenia within 1 week prior to study drug administration
* Patients must discontinue all herbal supplements at a minimum of one week prior to initiation of therapy (such information will be collected on each patient
* Requirement for routine use of hematopoietic growth factors (including granulocyte colony stimulating factor, granulocyte macrophage colony stimulating factor, or interleukin-11) or platelet transfusions to maintain absolute neutrophil counts or platelets counts above the required thresholds for study entry.
* Patient has an underlying, predisposing condition of bleeding or currently exhibits signs of bleeding. The subject has a recent history of non-chemotherapy induced thrombocytopenic associated bleeding within 1 year prior to the first dose of study drug.
* History or symptoms of cardiovascular disease (NYHA Class 2, 3, or 4; see Appendix B, New York Heart Association Criteria) within the last 6 months, particularly coronary artery disease, arrhythmias, or conduction defects with risk of cardiovascular instability, uncontrolled hypertension, clinically significant pericardial effusion, or congestive heart failure.
* Hypersensitivity to 4-aminoquinoline compounds, including hydroxychloroquine sulfate, chloroquine phosphate and amodiaquine.
* Prior history of treatment with ABT-263
* Known G-6PDH deficiency
* Retinal or visual field changes from prior 4-aminoquinoline compound use such as hydroxychloroquine sulfate, chloroquine phosphate and amodiaquine.
* Patients presenting with untreated cord compression are not eligible (patients with prior treatment and stability will be eligible)
* Concurrent use of other investigational agent
* Subject has undergone an allogeneic stem cell transplant
* Subject has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis
* Subject has a significant history of cardiovascular disease (e.g., MI, thrombotic or thromboembolic event in the last 6 months), renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic disease that in the opinion of the Investigator would adversely affect his/her participating in this study. Subject has received a biologic agent for anti-neoplastic intent within 30 days prior to the first dose of study drug.
* Subject is currently receiving or requires anticoagulation therapy (e.g., warfarin at any dose) or any drugs (e.g., aspirin, clopidogrel, etc) or herbal supplements that affect platelet function, with the exception of low molecular weight heparin or heparin that are used to maintain the patency of a catheter.
* Subject has received aspirin or warfarin within 7 days prior to the first dose of study drug.
* Subject has consumed grapefruit or grapefruit products within 3 days prior to the first dose of study drug.
* Received potent CYP3A inhibitors (e.g., ketoconazole) or inducers (substrates of CYP2D6) within 7 days prior to the first dose of study drug.
* Subject has received rifampin within 4 days prior to first dose of ABT-263

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert DiPaola, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey. The study was open to accrual on 6/4/2013 and was closed by the Principal Investigator on 3/3/2016 due to slow accrual.
Pre-assignment Details: We are reporting results on 13 eligible patients. Arm A dose escalation was completed. The study was then closed to due to slow accrual and the Investigator leaving the organization.
Groups:
- ARM A - Dose Escalation: Dose level 0: Abiraterone 1000 mg po daily and ABT-263 150 mg po daily Dose level 1: Abiraterone 1000 mg po daily and ABT-263 250 mg po daily* Dose level 2 (maximum planned phase II dose): Abiraterone 1000 mg po daily and ABT-263 350 mg po daily*
  * All patients at the 250 mg/day and 325 mg/day doses will start at 150 mg/day for the first 7 days (on Day -7) and escalated to their respective full dose on Day 1 if no DLT is observed and platelets are >50,000/mm3.
  NOTE: The dose escalation for ABT-263 combined with abiraterone was completed first prior to dose escalation with ABT-263 combined with hydroxychloroquine and abiraterone. Following both dose escalation portions of the trial, patients will then, and only then, be assigned to Arm A or Arm B of the phase II portion of the trial on a rotating basis of every other patient.
- ARM B - Dose Escalation: Dose level 0: Abiraterone 1000 mg po daily, ABT-263 150 mg po daily, Hydroxychloroquine 200 mg po BID daily Dose level 1: Abiraterone 1000 mg po daily and ABT-263 250 mg po daily*, Hydroxychloroquine 400 mg po BID daily Dose level 2 (maximum planned phase II dose): Abiraterone 1000 mg po daily and ABT-263 325 mg po daily*, Hydroxychloroquine 400 mg po BID daily
  * All patients at the 250 mg/day and 325 mg/day doses will start at 150 mg/day for the first 7 days (on Day -7) and escalated to their respective full dose on Day 1 if no DLT is observed and platelets are >50,000/mm3.
Period: Overall Study
Arm/Group | ARM A - Dose Escalation | ARM B - Dose Escalation
Started | 13 | 0
Completed | 13 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM A - Dose Escalation | ARM B - Dose Escalation | Total
Number analyzed (Participants) | 13 | 0 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 11 |  | 11
Age, Continuous [Median (Full Range); unit: years] | 69 [48 to 82] |  | 69 [48 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 |  | 0
  Male | 13 |  | 13
Region of Enrollment [Number; unit: participants]
  United States | 13 |  | 13

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Response to ABT-263 and Abiraterone and to ABT-263 in Combination With Hydroxychloroquine and Abiraterone in Patients That Are Progressing on Abiraterone
Description: Characterize "biochemical response" to ABT-263 and Abiraterone and to ABT-263 in combination with hydroxychloroquine and Abiraterone by looking at PSA levels.
Time Frame: 5 years
Population: Study was terminated early and insufficient data was collected to assess this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- ARM A: Abiraterone with ABT-263
  Abiraterone: ARM A and ARM B
  ABT-263: ARM A and ARM B
- ARM B: Abiraterone with both ABT-263 and Hydroxychloroquine
  Abiraterone: ARM A and ARM B
  ABT-263: ARM A and ARM B
  Hydroxychloroquine: ARM B
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 13 | 0
Participants | 0 |

2. Secondary Outcome: Time to PSA Progression
Time Frame: 5 years
Population: Study was terminated early and insufficient data were collected to assess this outcome measure.
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

3. Secondary Outcome: Progression Free Survival
Time Frame: 5 years
Population: Study was terminated early and insufficient data were collected to assess this outcome measure.
Arm/Group | ARM A - Dose Escalation | ARM B - Dose Escalation
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

4. Secondary Outcome: Measurable Tumor Response in Patients With Measurable Disease
Time Frame: 5 years
Population: Study was terminated early and insufficent data was collected to assess this outcome measure.
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

5. Secondary Outcome: Circulating Tumor Cells Pre-enrollment and During Therapy
Time Frame: 5 years
Population: Study was terminated early and insufficient data was collected to assess this outcome measure.
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

6. Secondary Outcome: Bcl-2 Family Protein Expression (Bcl-2, Bcl-XL, MCL-1) in Paraffin Blocks When Available by Immunohistochemistry
Time Frame: 5 years
Population: Study was terminated warly and insufficient data was collected to assess this outcome measure.
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

7. Secondary Outcome: Biomarkers of Autophagy Modulation by EM; and LC3, and/or p62 by Immunoblotting in PBMC and Tumor Tissue When Available
Time Frame: 5 years
Population: Study was terminated early and insufficient data was collected to assess this outcome measure.
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

8. Secondary Outcome: Overall Survival
Time Frame: 5 years
Population: Study was terminated early and insufficient data was collected to assess this outcome measure.
Arm/Group | ARM A | ARM B
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Arm/Group | ARM A - Dose Escalation | ARM B - Dose Escalation
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/0
Other Adverse Events (participants affected / at risk) | 13/13 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A - Dose Escalation (N=13) | ARM B - Dose Escalation (N=0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM A - Dose Escalation (N=13) | ARM B - Dose Escalation (N=0)
Nausea (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (13) | 0 (0)
Platelet count decreased (Investigations) | 11 (27) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (19) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (5) | 0 (0)
Fatigue (General disorders) | 8 (12) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 6 (9) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes